CLINICAL TRIAL: NCT06431438
Title: A Phase I Clinical Trial to Evaluate the Tolerability, Safety, Pharmacokinetics and Pharmacodynamics of TQA3810 Tablets
Brief Title: Study to Evaluate the Tolerability, Safety, Pharmacokinetics and Pharmacodynamics of TQA3810 Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: TQA3810-I-01
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- 0.5mg single-dose (Placebo Comparator): Ten subjects were enrolled, of whom 8 received the trial drug and 2 received placebo.
  Interventions: Drug: TQA3810
- 1.0mg single-dose (Placebo Comparator): Ten subjects were enrolled, of whom 8 received the trial drug and 2 received placebo.
  Interventions: Drug: TQA3810
- Food impact group (Other): Sixteen subjects were enrolled and all received the trial drug.
  Interventions: Drug: TQA3810
- 0.1mg single-dose (Placebo Comparator): Ten subjects were enrolled, of whom 8 received the trial drug and 2 received placebo.
  Interventions: Drug: TQA3810
- 0.3mg single-dose (Placebo Comparator): Ten subjects were enrolled, of whom 8 received the trial drug and 2 received placebo.
  Interventions: Drug: TQA3810
- Drug interaction group (Active Comparator): Sixteen subjects were enrolled and all received the trial drug.
  Interventions: Drug: TQA3810
- 0.1mg multiple dosing (Placebo Comparator): Ten subjects were enrolled, of whom 8 received the trial drug and 2 received placebo.
  Interventions: Drug: TQA3810
- 0.3mg multiple dosing (Placebo Comparator): Ten subjects were enrolled, of whom 8 received the trial drug and 2 received placebo.
  Interventions: Drug: TQA3810
- 0.5mg multiple dosing (Placebo Comparator): Ten subjects were enrolled, of whom 8 received the trial drug and 2 received placebo.
  Interventions: Drug: TQA3810
- 0.2mg multiple dosing (Placebo Comparator): Ten subjects were enrolled, of whom 8 received the trial drug and 2 received placebo.
  Interventions: Drug: TQA3810

INTERVENTIONS:
Drug: TQA3810 — TQA3810 is a small-molecule Toll-like receptor (TLR8) agonist

SUMMARY:
This study was a single-center study, including randomized, double-blind, placebo-controlled, single-dose escalation study, multiple-dose study, food effect on pharmacokinetics and drug metabolism transformation study, drug interaction study. To evaluate the tolerability, pharmacokinetics and metabolic transformation of TQA3810 in healthy subjects after single or multiple doses of TQA3810, the drug-drug interactions between TQA3810 tablets and entecavir dispersible tablets, and the pharmacokinetic properties of TQA3810 tablets in combination.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent before the trial, and fully understand the trial content, process and possible adverse reactions;
* Able to complete the study according to the requirements of the trial protocol;
* The participants (including their partners) are willing to voluntarily use effective contraceptive methods within 6 months from screening until the last dose of study drug, as detailed in the Appendix;
* Male and female subjects aged 18-55 years old (including 18 and 55 years old);
* The body weight of male subjects should not be less than 50 kg and the body weight of female subjects should not be less than 45 kg. Body mass index (BMI) = weight (kg)/height 2 (m2), BMI in the range of 18-28 kg/m2 (including the cut-off value);
* The physical examination and vital signs were normal or abnormal without clinical significance.

Exclusion Criteria:

* Smoking more than 5 cigarettes per day in the 3 months before the study;
* Allergic constitution (multi-drug and food allergy);
* A history of drug and/or alcohol abuse (drinking 14 units of alcohol per week: 1 unit = 285 mL beer, or 25 mL spirits, or 100 ml wine);
* Donation or massive blood loss (> 400 mL) within 3 months before screening;
* Taking any drugs that alter liver enzyme activity 28 days before screening;
* Have taken any prescription medication, over-the-counter medication, any vitamin product or herbal medicine within 14 days before screening;
* Those who had taken special diet (including dragon fruit, mango, grapefruit, etc.) or had strenuous exercise within 2 weeks before screening, or had other factors affecting drug absorption, distribution, metabolism, and excretion;
* Combined with the following inhibitors or inducers of CYP3A4, P-gp, or Bcrp, such as itraconazole, ketoconazole, or dronedarone, within three months before taking the study drug;
* A recent major change in diet or exercise habits;
* Have taken a study drug or participated in a clinical trial of the drug within three months before taking the study drug;
* A history of dysphagia or any gastrointestinal disorder affecting drug absorption or a history of cholecystectomy or biliary tract disease;
* Have any condition that increases the risk of bleeding, such as hemorrhoids, acute gastritis or gastric and duodenal ulcers;
* With severe systemic diseases and related medical history (including subjects with active or occult tuberculosis, a history of tuberculosis, or clinical manifestations suspected of tuberculosis), as well as immune system diseases and medical history;
* Had systemic or local infection within 2 months prior to screening, and were hospitalized for severe infection and/or required intravenous antibiotics;
* Subjects who were unable to tolerate a standard meal;
* An electrocardiogram (ECG) abnormalities have clinical significance;
* The female subjects were lactating or seropositive for pregnancy during the screening or test period;
* Clinically significant abnormalities on clinical examination or other clinical findings within 6 months prior to screening (including but not limited to gastrointestinal, renal, hepatic, neurological, hematologic, endocrine, oncologic, pulmonary, immune, psychiatric, or cardio-cerebrovascular diseases);
* Clinically significant fundus lesions (symptomatic cotton-like fundus changes) and retinopathy;
* Viral hepatitis (including hepatitis B and C), AIDS antibody, treponema pallidum antibody positive;
* From the screening stage to the onset of acute illness or concomitant medication before study medication;
* Consumption of chocolate, any caffeinated or xanthine-rich food or beverage 24 hours before taking the study drug;
* Have taken any alcohol-based product within 24 hours before taking the study medication;
* Having a positive urine drug screen or having a history of drug abuse or drug use in the past 5 years;
* Subjects with other factors considered by the investigator to be ineligible for the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 759 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | From the subject signed the informed consent form to 30 days after the last dose
  Occurrence of all adverse events (AEs), serious adverse events (SAEs), and treatment-related adverse events (TEAEs) were recorded.

SECONDARY OUTCOMES:
Cmax | Single dose escalation study: within 60 minutes pre-dose of day 1; 5, 10, 20, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 7, and 12 hours post-dose
  Maximum plasma drug concentration
Tmax | Single dose escalation study: within 60 minutes pre-dose of day 1; 5, 10, 20, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 7, and 12 hours post-dose
  To maximum plasma drug concentration time.
Half-life (t1/2) | Single dose escalation study: within 60 minutes pre-dose of day 1; 5, 10, 20, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 7, and 12 hours post-dose
  Drug half-life in plasma.
AUC0-t | Single dose escalation study: within 60 minutes pre-dose of day 1; 5, 10, 20, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 7, and 12 hours post-dose
  Plasma drug concentration from time 0 to the last measurable area under the drug concentration time curve.
AUC0-∞ | Single dose escalation study: within 60 minutes pre-dose of day 1; 5, 10, 20, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 7, and 12 hours post-dose
  Area under the plasma drug concentration time curve from time 0 to infinity.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital Affiliated to Medical School of Nanjing University, Nanjing, Jiangsu, China